CLINICAL TRIAL: NCT05570812
Title: In Vivo Targeting of Neuroactive Steroid and Immune Networks for Depression in People Living With HIV
Brief Title: Neuroactive Steroid to Treat Depressed Mood: A Trial for People With HIV
Acronym: SOOTHE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Institute for Medical Research, Inc. (Other)
Responsible Party: Principal Investigator, Shibani Mukerji, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P001941; 1R01MH131194-01 (NIH)
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Anxiety Depression; HIV
Keywords: HIV; Depression; Neuroactive Steroid; Pregnenolone
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pregnenolone; Neurosteroids

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive oral pregnenolone or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled trial. All roles will be masked except the research pharmacist and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Experimental): Participants will be on the following dosage schedule:
  50 mg daily for 2 weeks, THEN 100 mg daily for 1 week, THEN 250 mg daily for 1 week, THEN 500 mg daily for 4 weeks
  Interventions: Drug: Placebo
- Pregnenolone (Experimental): Participants will be on the following dosage schedule:
  50 mg daily for 2 weeks, THEN 100 mg daily for 1 week, THEN 250 mg daily for 1 week, THEN 500 mg daily for 4 weeks
  Interventions: Drug: Pregnenolone

INTERVENTIONS:
Drug: Placebo — (4-week ramp, 4-week steady dosing)
  Arms: Placebo
Drug: Pregnenolone — (4-week ramp, 4-week steady dosing)
  Other Names: Neuroactive steroid
  Arms: Pregnenolone

SUMMARY:
This study will determine the effects of pregnenolone on brain function, inflammation and depressive symptoms in people with HIV who have depression. Participants in this study will receive a pill of either pregnenolone or placebo, and can stay on their current antidepression medications. Brain imaging and behavioral assessments will be performed during the study.

DETAILED DESCRIPTION:
Pregnenolone is a neuroactive steroid that exhibits actions highly relevant to treating depression in people with HIV. The investigators' recent human data suggest that neuroactive steroids are decreased in people with HIV and depression. In addition, multiple groups have reported reductions in neuroactive steroids in people without HIV who have depression. A total of 120 people living with HIV on antiretroviral therapy with depression will be randomized to either pregnenolone or placebo (2 groups/90 participants receiving pregnenolone and 30 participants receiving placebo). Drug dosage will begin at 50 mg daily and incrementally increase to 500 mg daily within the first 4 weeks, with a stable 500 mg/day regimen for the final 4 weeks. Behavioral testing and blood draw will be performed at baseline, 2 weeks, 4 weeks, and 8 weeks, while magnetic resonance spectroscopy (MRS), and task-based functional magnetic resonance imaging (MRI) will be conducted at 2 weeks and 8 weeks.

The investigators hypothesize that pregnenolone will be well-tolerated in people with HIV and depression, and that this intervention may improve brain activity and reduce inflammation.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years
* HIV-1 viral load <200 copies/mL on antiretroviral therapy (ART) at screening visit
* Center for Epidemiological Studies - Depression (CES-D) score ≥ 20

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI) or poor-quality baseline MRI preventing image analyses as determined by radiologist assessment
* Recent severe infections including opportunistic infections, active bacterial, mycobacterial, fungal, or certain viral infections
* Vulnerable populations (e.g., pregnant/nursing, severe cognitive or intellectual impairment, incarcerated)
* Use of cobicistat or ritonavir
* High risk for suicide (active suicidal ideation (SI) with plan/intent as assessed by using the Columbia Suicide Severity Rating (C-SSRS) or > 2 attempts in lifetime or any in the past 6 months) or expresses homicidal ideation necessitating clinical intervention or representing an imminent concern
* Any severe (life-threatening or unstable) medical condition as determined by clinician assessment
* Blood pressure, with the lowest reading taken after three repeat readings during screening visit, ≥ 160 mmHg systolic OR ≥ 95 mmHg diastolic or other life-threatening vital signs as determined by clinician assessment
* Clinically significant abnormalities in physical examination or ECG that would interfere with study participation
* Decompensated cirrhosis, active liver inflammation (alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥ 5 times the upper limit of normal) or unsuppressed viral hepatitis B or C infection
* Severe renal disease (estimated glomerular filtration rate ≤ 30 mL/min/1.73m2)
* Seizure disorder requiring antiepileptic treatment
* History of allergic reaction or side effects with prior pregnenolone use
* Currently using testosterone enanthate, testosterone cypionate, or estrogen containing preparations that significantly increase systemic estrogen levels, including but not limited to oral and transdermal forms of estrogen. All other forms of exogenous sex steroid hormones will be evaluated at the discretion of the PI and/or clinical delegates.
* Currently using systemic immunosuppressive agents, including corticosteroids, chemotherapy, or specific immunomodulating agents, such as monoclonal antibodies and TNF-inhibitors
* Excessive alcohol or other substances use that would interfere with classification of major depression disorder, study procedures and/or follow-up
* Current diagnosis of bipolar disorder
* Diagnosis of a psychotic disorder (current or lifetime)
* Diagnosis of schizophrenia (current or lifetime)
* <70% adherence to study drug prior to randomization
* Inability to swallow pills/capsules
* Not able to complete neuropsychological testing in English
* Concurrent participation in another interventional trial, except for lifestyle and device studies (For vaccination studies, individuals in the observation period are not exclusionary. Other interventions will be evaluated at the discretion of the PI and/or clinical delegates.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Gamma-aminobutyric acid (GABA) Concentration | Day 14, Day 56
  Comparison between Pregnenolone and Placebo Groups of Left Insular Cortex GABA Concentration, Adjusted for Baseline.

SECONDARY OUTCOMES:
Center for Epidemiological Studies-Depression (CES-D; scores range from 0 (no symptoms) to 60 (maximum severity of depressive symptoms)) | Day 0, Day 14, Day 56
  Comparison of Percentage of Pregnenolone and Placebo Groups Showing Clinical Improvement of Depression at Study End. The revised CES-D is administered, and the total score is calculated by adding the responses to the 20 questions.
CD14+CD16+ Monocytes | Day 0, Day 14, Day 28, Day 56
  Comparison of the Percentage of CD14+CD16+ Monocytes Over Time Adjusted for Baseline Between Pregnenolone and Placebo Groups
GABA Concentration in Responders | Day 0, Day 14, Day 56
  Comparison of Baseline Left Insular Cortex GABA and Pregnenolone Between Participants in Pregnenolone Group with Clinical Improvement Compared to Clinical Non-Improvers in Pregnenolone Group
Adverse Events | Day 14, Day 56
  Comparison of the Incidence and Severity of Adverse Events Between Pregnenolone and Placebo Groups
Dose Modifications | Day 14, Day 56
  Comparison of Dose Modifications Required Between Pregnenolone and Placebo Groups

CONTACTS AND LOCATIONS:
Overall Officials: Shibani S. Mukerji, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mukerji SS, Misra V, Lorenz DR, Chettimada S, Keller K, Letendre S, Ellis RJ, Morgello S, Parker RA, Gabuzda D. Low Neuroactive Steroids Identifies a Biological Subtype of Depression in Adults with Human Immunodeficiency Virus on Suppressive Antiretroviral Therapy. J Infect Dis. 2021 May 20;223(9):1601-1611. doi: 10.1093/infdis/jiaa104. PMID 32157292